CLINICAL TRIAL: NCT01891812
Title: Nitrous Oxide for Analgesia in Sickle Cell Vaso-occlusive Crisis
Brief Title: Nitrous Oxide Analgesia Vaso-occlusive Crisis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel S Tsze, MD, MPH, Associate Professor of Pediatrics in Emergency Medicine, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAK6900
Record Dates: First submitted 2013-06-29; First posted 2013-07-03 (Estimated); Results first posted 2024-07-16 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sickle Cell Disease; Vaso-occlusive Crisis
Keywords: Sickle cell disease; Vaso-occlusive crisis; Nitrous oxide; Emergency department
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Nitrous oxide 50% (Experimental): Nitrous oxide 50% administered for 20 minutes.
  Interventions: Drug: Nitrous oxide 50%

INTERVENTIONS:
Drug: Nitrous oxide 50%

SUMMARY:
Patients who have sickle cell VOC are usually treated with opioids, such as morphine. However, this current way of treating them has not improved the health, medical outcomes, or rates of hospitalizations. In addition, since VOC can happen very frequently over a long period of time, giving opioids over and over again can cause both short-term and long-term problems. Nitrous oxide (N2O) is a way of treating pain that may provide a better alternative to repeatedly giving opioids over long periods of time. N2O has been shown to provide up to 3 hours of pain relief in inpatient patients with VOC whose pain did not improve with morphine infusions, and is used extensively in France, where almost half of 85 pediatric emergency departments use nitrous oxide to treat children with VOC whose pain did not get better with standard treatment with morphine. However, pain relief which N2O provides in the acute setting has not been well described. Therefore, the purpose of our study is to describe how well N2O can relieve the pain in patients with SCD who present to the emergency department and are experiencing a VOC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sickle cell disease
* Ages 8 to 18, inclusive
* Present to the pediatric emergency department with VOC and whose pain scores remain greater than or equal to 7/10 on the NRS after initial standard treatment (i.e. IV fluids, morphine and NSAIDs).

Exclusion Criteria:

* life-threatening illness as determined by attending clinician
* developmental delay
* altered level of consciousness
* any contraindications to receiving N2O
* foster children and wards of the state

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2013-11-12 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Tsze, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- New York Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States

REFERENCES:
- [Result] Tsze DS, Licursi M, Ender KL, Kennedy RM, Dayan PS. Nitrous Oxide for Treating Vaso-Occlusive Crisis Pain in Children With Sickle Cell Disease: A Pilot Study. Acad Emerg Med. 2025 Nov 28. doi: 10.1111/acem.70203. Online ahead of print. No abstract available. PMID 41315052

RESULTS

PARTICIPANT FLOW:
Groups:
- Nitrous Oxide: Patients with Sickle cell disease and experiencing vaso-occlusive crises (VOC) with a pain score of greater than or equal to 7/10.
  Patients will receive the standard care of IV fluids, NSAIDs, and IV morphine or hydromorphone. The pain score will be reassessed 15 minutes after the initial pain scoring, and if the pain score is still greater than or equal to 7/10, nitrous oxide (N2O) will be administered at a concentration of 50% for 20 minutes.
Period: Overall Study
Arm/Group | Nitrous Oxide
Started | 5
Completed | 0
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  0 - 7 years | 0
  8 - 17 years | 5
  18 - 65 years | 0
  >65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 0
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Patient-reported pain score immediately after administration of nitrous oxide. The full range of the pain score is 0 to 10; 0 = no pain, 10 = worst pain.
Time Frame: Up to 4 hours
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 5
score on a scale | 5.7 [4.6 to 6.8]

2. Secondary Outcome: Duration of Analgesia
Description: Duration of analgesia (minutes) from time of administration of nitrous oxide until administration of additional analgesia.
Time Frame: Up to 4 hours
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 5
minutes | 39 [16 to 60]

3. Other Pre Specified Outcome: Number of Participants With Peripheral Neuropathies
Description: Complaints or physical ﬁndings suggestive of peripheral neuropathies (which may present as numbness, tingling, pain, or loss of feeling in ﬁngers or toes; or weakness or difﬁculty moving the arms or legs) at the 8 week follow-up
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 5
Participants | 0

4. Other Pre Specified Outcome: Number of Participants With Macrocytic Anemia
Description: The presence of macrocytic anemia at 8 weeks time in patients who had low vitamin B12 levels at the time of enrollment.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Nitrous Oxide
Number analyzed (Participants) | 5
Participants | 0

ADVERSE EVENTS:
Time Frame: Up to 4 hours
Arm/Group | Nitrous Oxide
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 2/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nitrous Oxide (N=5)
Nausea (General disorders) | 1
Vomiting (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT01891812/Prot_SAP_000.pdf